CLINICAL TRIAL: NCT01938716
Title: Tissue Pharmacokinetics of Intraoperative Gemcitabine in Adenocarcinoma of the Pancreas After Preoperative Chemoradiation Therapy
Brief Title: Gemcitabine Pharmacokinetics After Preoperative Chemoradiation Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early termination due to low accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-0703; NCI-2013-02211 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Results first posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Adenocarcinoma of the Pancreas; Intratumoral gemcitabine levels; Pancreatic surgery; Pharmacokinetic testing; PK; Gemcitabine; Gemcitabine Hydrochloride; Gemzar
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gemcitabine Infusion (Experimental): Gemcitabine administered intravenously as a dose of 500 mg/m2 at a fixed dose rate of 10 mg/m2/min for the first 5 patients (to validate hematologic safety). Next 15 subsequent patients receive 750 mg/m2 at a fixed dose rate of 10 mg/m2/min. The drug infusion started 50-75 minutes prior to complete gross tumor removal (timing dependent on dose) in order to have drug administration complete at tumor removal.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — 500 mg/m2 at a fixed dose rate of 10 mg/m2/min by vein for the first 5 patients during pancreatic surgery. Next 15 subsequent patients receive 750 mg/m2 by vein at a fixed dose rate of 10 mg/m2/min.
  Other Names: Gemcitabine Hydrochloride; Gemzar

SUMMARY:
The goal of this clinical research study is to learn if gemcitabine given during surgery can enter pancreas cancer cells in patients who have already received chemotherapy and radiation.

Gemcitabine is a drug used to treat pancreatic cancer. However, it has not previously been studied if gemcitabine can enter pancreatic cancer cells. Gemcitabine is designed to block the growth of cancer cells, which may cause cancer cells to die.

DETAILED DESCRIPTION:
Surgery:

If you agree to take part in this study, your surgery will be performed in the same way as it would be even if you were not taking part in this study. You will sign a separate consent form for surgery. The length of the surgery and the time you are under anesthesia will not be changed by taking part in the study.

During surgery, you will have routine procedures to learn if the disease has spread to other areas. If the disease has spread beyond the pancreas, surgical removal will not be possible.

If there are no signs of spread or other reasons the cancer cannot be removed, the surgeon will begin the process of removing the disease.

Study Drug Administration:

You will receive gemcitabine by vein during surgery. Gemcitabine will be given through an infusion catheter that is placed in your arm or chest in the operating room after you are asleep.

The infusion catheter is a standard-of-care procedure for all participants who are having this surgery. You will be asked to sign a separate consent form for the infusion catheter.

The infusion will take either 50 or 75 minutes, depending upon when you joined the study. The first 5 participants will receive gemcitabine over 50 minutes and the rest of the participants will receive gemcitabine over 75 minutes.

Blood and Tissue Collection:

Up to 8 blood samples (about 1 tablespoon each time) will be drawn over 70-95 minutes for pharmacokinetic (PK) testing on the day of surgery. PK testing measures the levels of study drug in your blood at different time points. The blood will also be used for biomarker testing. Biomarkers are chemical markers found in the blood and tissue that may be related to your reaction to the study drug.

Some of the tumor tissue and normal tissue removed during surgery will be collected to learn if gemcitabine is able to enter the tissue cells and for biomarker testing.

Length of Participation:

If for any reason during the surgery the surgeon decides that removal of the pancreas is not possible, you will not receive gemcitabine and your participation in this study will end.

Your active participation in this study will be over once you have had surgery and completed the follow-up.

Follow-Up:

One (1) time each day while you are in the hospital recovering from the surgery and then at the time of a routine clinic visit or by phone call at least 1 time a week, for up to 30 days after surgery, you will be asked if you have had any side effects.

This is an investigational study. Gemcitabine is FDA approved and commercially available for the treatment of pancreatic cancer. Its use during surgery is investigational.

Up to 40 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologic or histologic proof of adenocarcinoma of the pancreas is required. Patients with Islet cell tumors are not eligible.
2. Patients do not have known metastases.
3. Patients must have potentially resectable or borderline resectable pancreatic cancer and have agreed to undergo surgical resection at MD Anderson Cancer Center if operable. They will have undergone staging (physical examination, chest x-ray, contrast enhanced CT or MRI (if CT contraindicated) and/or angiogram) to determine resectability.
4. Patients have completed radiation and chemotherapy with either fluoropyrimidines (5-FU or capecitabine) or gemcitabine as a radiosensitizing agent as part of their preoperative therapy. Previous systemic chemotherapy alone is not allowed. Preoperative therapy will be completed at least 4 weeks prior to surgery.
5. Patients with Karnofsky performance status > 70 are eligible.
6. There will be no upper age restriction. Patients less than 18 years of age are excluded from the protocol because adenocarcinoma of the pancreas is rarely seen in the pediatric population.
7. Adequate renal and bone marrow function: Leukocytes >= 3,000/uL; Absolute neutrophil count >= 1,500/uL; Platelets >= 100,000/Ul; Serum creatinine <= 2.0 mg/dL; Creatinine clearance >= 60 ml/min (calculated by the Cockcroft -Gault equation)
8. Adequate Hepatic function (endoscopic or percutaneous drainage as needed): Total bilirubin < = 3 X institutional upper limits of normal (ULN); AST (SGOT)/ALT (SGPT) <= 5 X institutional ULN
9. Patients must have no fever or evidence of infection or other coexisting medical condition that would preclude administration of gemcitabine. Patients with uncontrolled congestive heart failure, unstable angina and myocardial infarction within 3 months will be excluded.
10. Patient is not pregnant. Women of childbearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use acceptable contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) and refrain from breast-feeding, as specified in the informed consent.
11. Patients must sign a study-specific consent form.

Exclusion Criteria:

1. Major cardiovascular or pulmonary comorbidity that precludes use of general anesthesia (NYHA [New York Heart Association] Class III and IV).
2. Identification of metastatic disease.
3. Patients with a known hypersensitivity to Gemcitabine.
4. Pregnant women
5. Inability to comply with study and/or follow-up procedures.
6. Patients < 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gauri Varadhachary, MD, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: March 2012 to February 2015. All recruitment done at The University of Texas, MD Anderson Cancer Center.
Groups:
- Intraoperative Gemcitabine Administration: Gemcitabine administered intravenously at dose of 500 - 750 mg/m2 at a fixed dose rate of 10mg/m2/min, 50-75 minutes prior to complete gross tumor removal.
Period: Overall Study
Arm/Group | Intraoperative Gemcitabine Administration
Started | 12
Completed | 8
Not Completed | 4
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intraoperative Gemcitabine Administration
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: To Quantifiably Assess Intratumoral Gemcitabine Levels in Human Pancreatic Cancer Tissue After a Single Intraoperative Infusion in Patients.
Description: The quantification of serum, PBMC, and cancer tissue levels of gemcitabine from frozen samples will be assessed using standardized techniques in high performance liquid chromatography-mass spectometry (HPLC/MS).
Time Frame: through study completion, up to 2 years and 6 months
Population: Samples inadequate for testing to meet objective; early termination of protocol due to low accrual.
Arm/Group | Intraoperative Gemcitabine Administration
Number analyzed (Participants) | 0

2. Secondary Outcome: To Measure Intra-DNA Gemcitabine (dFdC) Levels Using a Novel Assay Liquid Chromatography-mass Spectometry (LC/MS/MS).
Description: Gemcitabine incorporation in DNA will be quantified by a proprietary LC/MS/MS method developed by Eli Lilly and performed by Advion BioServices. DNA extracted from the tissue samples to be sent to Advion.
Time Frame: through study completion, up to 2 years and 6 months
Population: Samples inadequate for testing to meet objective; early termination of protocol due to low accrual.
Arm/Group | Intraoperative Gemcitabine Administration
Number analyzed (Participants) | 0

3. Secondary Outcome: To Assess and Validate Previously Described Markers That May be Predictive of Gemcitabine Sensitivity or Resistance.
Description: The mRNA level is measured using real time PCR and protein expressed by IHC, Gene expression level will be correlated to the gemcitabine measurements. Additionally measure markers of proliferation and apoptosis by p21and ki67 IHC and fluorescent TUNEL analysis.
Time Frame: through study completion, up to 2 years and 6 months
Population: Samples inadequate for testing to meet objective; early termination of protocol due to low accrual
Arm/Group | Intraoperative Gemcitabine Administration
Number analyzed (Participants) | 0

4. Secondary Outcome: To Measure the Impact of Microvessel Density and the Molecular Expression Level of the Hh Signaling Pathway on Gemcitabine Delivery and DNA Incorporation.
Description: The mRNA and protein expression of SHH, Gli, and SMO will be measured by RT-PCR and IHC method, respectively.
Time Frame: through study completion, up to 2 years and 6 months
Population: Samples inadequate for testing to meet objective; early termination of protocol due to low accrual.
Arm/Group | Intraoperative Gemcitabine Administration
Number analyzed (Participants) | 0

5. Secondary Outcome: To Correlate Intratumoral Gemcitabine Levels and Its Tumoricidal Activity With Ki67 Index and Intratumoral Apoptosis.
Description: Measure markers of of proliferation and apoptosis by p21 and ki67 IHC and fluorescent TUNEL analysis.
Time Frame: through study completion, up to 2 years and 6 months
Population: Samples inadequate for testing to meet objective; early termination of protocol due to low accrual.
Arm/Group | Intraoperative Gemcitabine Administration
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data collected from intraoperative gemcitabine infusion, during post-surgery hospitalization and followed for 30 day post surgery
Arm/Group | Intraoperative Gemcitabine Administration
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intraoperative Gemcitabine Administration (N=8)
White blood cell decreased (Investigations) | 5
Anemia (Blood and lymphatic system disorders) | 1
Neutrophilcount decreased (Investigations) | 3
Platelet count decreased (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-08-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT01938716/Prot_SAP_000.pdf